CLINICAL TRIAL: NCT00425477
Title: A Phase II Study of Bexarotene + Sargromastastin as Agents of Differentiation in MDS and AML
Brief Title: Bexarotene and GM-CSF in Treating Patients With Myelodysplastic Syndrome or Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0675 CDR0000525989; P30CA006973 (NIH); JHOC-J0675; JHOC-NA_00003076
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Results first posted 2018-09-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-09

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: refractory anemia with excess blasts; recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative disease, unclassifiable; refractory anemia with ringed sideroblasts; refractory cytopenia with multilineage dysplasia; chronic myelomonocytic leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult pure erythroid leukemia (M6b); adult erythroleukemia (M6a); adult acute megakaryoblastic leukemia (M7); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with inv(16)(p13;q22)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Acute; Myeloproliferative Disorders; Leukemia, Myelomonocytic, Chronic; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — sargramostim; Bexarotene; Cytogenetic Analysis; In Situ Hybridization, Fluorescence; Flow Cytometry; Biopsy

ARMS (1):
- Bexarotene + GM-CSF (Experimental): BEX and GM-CSF were administered in 4 week cycles. BEX was given orally with food daily for 28 days at the FDA-approved dose for treatment of CTCL of 300 mg/m2 and GM-CSF was given at a daily dose of 125 µg/m2 subcutaneously for 28 days.
  Interventions: Biological: sargramostim; Drug: bexarotene; Genetic: cytogenetic analysis; Genetic: fluorescence in situ hybridization; Other: flow cytometry; Other: laboratory biomarker analysis; Procedure: biopsy

INTERVENTIONS:
Biological: sargramostim
Drug: bexarotene
Genetic: cytogenetic analysis
Genetic: fluorescence in situ hybridization
Other: flow cytometry
Other: laboratory biomarker analysis
Procedure: biopsy

SUMMARY:
RATIONALE: Bexarotene may help cancer or abnormal cells become more like normal cells, and to grow and spread more slowly. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood. Giving bexarotene together with GM-CSF may be an effective treatment for myelodysplastic syndrome (MDS) or acute myeloid leukemia.

PURPOSE: This phase II trial is studying how well giving bexarotene together with GM-CSF works in treating patients with MDS or acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the clinical response in patients with myelodysplastic syndromes or acute myeloid leukemia treated with bexarotene and sargramostim (GM-CSF).

Secondary

* Determine the clinical activity of this regimen, in terms of transfusion requirements, in these patients.
* Determine the biological activity of this regimen, in terms of biological markers and cytogenetic abnormalities, in these patients.
* Assess the toxicity profile of this regimen in these patients.

OUTLINE: Patients receive oral bexarotene and sargramostim (GM-CSF) subcutaneously on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Blood and bone marrow samples are collected at baseline and after 1 or 2 courses of study therapy. Samples are examined by flow cytometry for laboratory studies, including biological markers, and by fluorescent in situ hybridization (FISH) for cytogenetic changes.

After completion of study treatment, patients are followed periodically for 6 months.

PROJECTED ACCRUAL: A total of 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis (confirmed by bone marrow aspirate and/or biopsy) of 1 of the following:

  * Myelodysplastic syndromes of 1 of the following cell types:

    * Refractory anemia (RA) with ringed sideroblasts
    * Refractory cytopenia with multilineage dysplasia (RCMD)
    * RCMD and ringed sideroblasts
    * RA with excess blasts-1
    * RA with excess blasts-2
    * Myelodysplastic syndromes, unclassified
    * Chronic myelomonocytic leukemia
  * Relapsed or refractory acute myeloid leukemia (AML), meeting 1 of the following criteria:

    * Recurrent genetic abnormalities (11q23 [MLL] abnormalities)
    * Multilineage dysplasia
    * Therapy-related AML
    * Not otherwise categorized, including any of the following:

      * M0 minimally differentiated
      * M1 without maturation
      * M2 with maturation
      * M4 myelomonocytic leukemia
      * M5 monoblastic/monocytic leukemia
      * M6 erythroid leukemia
      * M7 megakaryoblastic leukemia
* Newly diagnosed untreated AML allowed provided patient does not qualify for or refused potentially curative intensive chemotherapeutic regimens
* No RA with 5q-syndrome
* No peripheral leukemia with blast count > 30,000/mm³ (uncontrolled with hydroxyurea)
* Relatively stable bone marrow function for > 7 days (i.e., no WBC doubling to > 10,000/mm^3)
* No acute promyelocytic leukemia
* No clinical symptoms of active CNS disease (if CNS disease is suspected, patient must have lumbar puncture with negative cytology)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 1.6 mg/dL (unless secondary to hemolysis)
* AST and ALT ≤ 4 times upper limit of normal (unless disease related)
* Hemoglobin ≥ 8 g/dL (transfusions allowed)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No untreated positive blood cultures or progressive infection as assessed by radiographic studies
* No history of intolerance to sargramostim (GM-CSF)

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* At least 2 weeks since prior treatment for myeloid disorder, including any of the following:

  * Chemotherapy
  * Hematopoietic growth factors
  * Biologic therapy (e.g., monoclonal antibodies)
* Hydroxyurea for patients with WBC > 10,000/mm^3 allowed
* No concurrent vitamin A supplementation
* No concurrent gemfibrozil

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. Douglas Smith, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bexarotene + GM-CSF
Started | 26
Completed | 13
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Bexarotene + GM-CSF
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 72 [49 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response (Complete and Partial)
Description: Response to treatment was assessed after two cycles, according to International Working Group (IWG) criteria.
Time Frame: assessed after 2 cycles, up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bexarotene + GM-CSF
Number analyzed (Participants) | 13
Participants
  PR (partial remission) | 0
  HI (hematologic improvement) | 4
  SD (stable disease) | 4
  PD (progressive disease) | 5

2. Secondary Outcome: Clinical Activity as Measured by Change in Peripheral Blood Counts and Changes in Transfusion Requirements
Description: ANC count at baseline and after two cycles were measured and compared. Due to the limited number of clinical responders, the changes in transfusion requirements were not measured.
Time Frame: Baseline and after two cycles
Measure: Mean (Standard Error); unit: neutrophils/mm^3
Arm/Group | Bexarotene + GM-CSF
Number analyzed (Participants) | 13
neutrophils/mm^3
  ANC at baseline | 524 (95)
  ANC after 2 cycles | 931 (244)

3. Secondary Outcome: Biological Activity as Measured by in Vivo Induction of Terminal Differentiation of Myeloid Progenitors and in Vivo Changes in Detectable Chromosomal Abnormalities
Time Frame: Baseline and 6, 12, 24, and 36 weeks
Population: Due to the limited number of clinical responders, this research assay was not done.
Arm/Group | Bexarotene + GM-CSF
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Bexarotene + GM-CSF
All-Cause Mortality (participants affected / at risk) | 3/26
Serious Adverse Events (participants affected / at risk) | 7/26
Other Adverse Events (participants affected / at risk) | 7/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bexarotene + GM-CSF (N=26)
Neutropenic infection (Infections and infestations) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Atrial flutter (Cardiac disorders) | 1
acute subdural hemmorrhage (Nervous system disorders) | 1
sepsis (Blood and lymphatic system disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bexarotene + GM-CSF (N=26)
Elevated ALT (Hepatobiliary disorders) | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes